CLINICAL TRIAL: NCT04139265
Title: Accordance Between Transferrin Saturation Coefficient and Ferritinemia in Diagnosis of Iron Deficiency, in Patients Hospitalised in Internal Medicine Service and 65 Years Old and More
Brief Title: Transferrin Saturation Coefficient and Ferritinemia in Diagnosis of Iron Deficiency
Acronym: CarenceMartial
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0079
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Iron-deficiency; Internal Medicine; Transferrin; Ferritinemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized patients aged 65 and over: - Patients aged 65 and over hospitalized in the department of Internal Medicine and Geriatry
  Interventions: Diagnostic Test: biologic analysis (ferritinemia, transferrin saturation coefficient)

INTERVENTIONS:
Diagnostic Test: biologic analysis (ferritinemia, transferrin saturation coefficient) — Each patient will follow a blood test in order to compare between ferritinemia and transferrin saturation coefficient in iron deficiency diagnosis

SUMMARY:
Transferrin saturation coefficient and ferritinemia in diagnosis of iron deficiency

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years old
* Patient hospitalized in the internal medicine and geriatry service
* Patient affiliated with a social security scheme
* Patient signed an Informed consent

Exclusion Criteria:

* Risk benefit balance not in favor of iron deficiency check-up
* Patient in palliative care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly people hospitalized in the internal medicine and geriatry service
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Agreement between Transferrin Saturation Coefficient (TSC) and ferritinemia dosage | Day one
  The overall agreement, assessed by kappa Cohen

SECONDARY OUTCOMES:
Prevalence of iron deficiency with and without anaemia | Day one
  Number of patients with iron deficiency with or without anaemia
Prevalence of etiologies of iron deficiency | Day one
  Number of patients for each etiology
Prevalence of iron deficiency in patients with anticoagulant and platelet aggregation inhibitor | Day one

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Bulckaen, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille
Locations (1):
- Saint-Philibert hospital, Lomme, Nord, France

IPD SHARING:
Plan to Share IPD: No